CLINICAL TRIAL: NCT03053583
Title: Comparison of the Vocal Cord Views Using the Classical Miller, Wis-Hipple and C-MAC Straight Size 1 Blades in Young Children
Brief Title: Vocal Cord Views With the Classical Miller, Wis-Hipple and C-MAC Size 1 Blades in Young Children
Acronym: POGO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jerrold Lerman, Clinical Professor of Anesthesia, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Laryngoscopy2
Record Dates: First submitted 2014-11-19; First posted 2017-02-15 (Actual); Results first posted 2025-04-15 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-03

CONDITIONS: Percent of Vocal Cords (Glottic) Opening
Keywords: larynx, laryngoscopy; vocal cords, laryngoscopy; airway; pediatric
MeSH Terms: conditions — Laryngeal Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Miller Laryngoscope blade (Active Comparator): A photo of the best vocal cord view will be taken during laryngoscopy using Miller blade. The view of the vocal cords will be assessed using the POGO score by a blinded assessor.
  Interventions: Device: Laryngoscope blade
- Wis-Hipple Laryngoscope blade (Active Comparator): A photo of the best vocal cord view will be taken during laryngoscopy using Wis- Hipple blade. The view of the vocal cords will be assessed using the POGO score by a blinded assessor.
  Interventions: Device: Laryngoscope blade
- C-Mac Laryngoscope blade (Active Comparator): An image of the best vocal cord view will be saved on C-MAC monitor's SD card during laryngoscopy using C-MAC straight blade. The view of the vocal cords will be assessed using the POGO score by a blinded assessor.
  Interventions: Device: Laryngoscope blade

INTERVENTIONS:
Device: Laryngoscope blade — The POGO score assesses the percent of the glottic opening that can be seen with each blade
  Other Names: Miller laryngoscope blade; Wis- Hipple laryngoscope blade; C-MAC straight laryngoscope blade

SUMMARY:
The purpose of this study is to compare straight blades in obtaining best vocal cord view in children. The investigators will compare size 1 Classical Miller, size 1 Wis-Hipple, and size 1 C-MAC straight blades in young children.

DETAILED DESCRIPTION:
This will be a prospective, randomized, blinded study. The primary objective is to compare straight blades in obtaining best vocal cord view in children. The secondary objectives will be to determine the subjective ease of laryngoscopy and intubation, desaturation and complications with each blade and to compare the view of the CMAC with a photo of the direct view with the CMAC blade.

In this study, the investigators will compare three different straight blades used in pediatric anesthesia: Miller blade size 1, Wis-Hipple blade size 1, and C-MAC straight blade size 1.

The sample size was estimated in this equivalence study assuming an alpha two-tailed of 0.05, beta of 0.2, proportion with a POGO score > 80 with the Miller blade (based on the results of our previous study) of 0.64 and an estimated proportion of 0.74 with the Wis-Hipple blade in the present study. The hypothesized difference required to reject equivalence is ≥ 0.2. This requires 96 children in total or 32 children per group. To account for un-interpretable photos and dropouts, we enrolled 101 children.

One hundred and one children who were eligible to participate will be consented, randomized, and allocated to one of the three study groups after consent is obtained from the parents/ guardian during regular anesthesia pre-operative evaluation. According to randomization children will be assigned to one of three groups:

Group A- Laryngoscopy by classical Miller blade, size 1 Group B- Laryngoscopy by Wis-Hipple blade, size 1 Group C- Laryngoscopy by C-MAC Miller blade, size 1.

After induction of general anesthesia, the anesthesiologist will perform either direct laryngoscopy using the Classical Miller, Wis-Hipple or C-MAC blade or indirect laryngoscopy using the C-MAC video straight blade. Photography of the best vocal cord view will be taken during direct laryngoscopy and the image of best vocal cord view will be saved by C-MAC. At the conclusion of the study, the photographs from all 96 patients will be converted such that the quality of the images standardized using Adobe Photoshop will appear similar to two blinded anesthesiologists who are also unaware of the study hypothesis.

Recruitment Procedure There will not be recruitment in advance. During the pre-anesthesia assessment of the patients who need to undergo a surgery under general anesthesia they will be screened for the inclusion and exclusion criteria for the study. The parents/ guardian will be informed about the study, its objectives, purpose, risks and benefits.

Consenting Procedure The consent to participate in this study will be obtained from parents/ guardian during pre-anesthesia assessment of the child in the holding area. Privacy and confidentiality will be assured.

Randomization Procedure After obtaining consent each child will be assigned a random serial number. Randomization will be prepared using random number table by a person not involved in the study before the study begins. Accordingly the patient will be allocated to a study group depending upon the matching number.

Research Procedure

1. Induction of General anesthesia ASA standard monitors will be applied prior to induction of anesthesia. General anesthesia in all children will be induced by face mask using 70% N20 in O2 and 8% Sevoflurane at fresh gas flow 8 L/min. After loss of eyelash reflex a peripheral intravenous catheter will be placed. Propofol 2-3 mg/kg and Rocuronium 0.5 mg/kg will be given. After achievement of adequate anesthesia depth and preoxygenation laryngoscopy will be performed.
2. Laryngoscopy and Photography The laryngoscopy technique will be chosen according to randomization. In "group A" anesthesiologist will use size 1 classical Miller blade for direct laryngoscopy. The blade will be placed under epiglottis and a photo will be taken by a second anesthesiologist using a high-quality digital camera after obtaining best glottic view. Then tracheal intubation will be performed. In "group B" size 1 Wis-Hipple blade will be used for direct laryngoscopy in the same manner. In "group C" a size 1 C-MAC straight blade for indirect videolaryngoscopy will be used. The blade will also be placed under the epiglottis and a photo of the direct view with the C-MAC will be taken. In group C the second anesthesiologist will save the images of best vocal cord view on a SD card in the C-MAC monitor.

   The oxygen saturation, blood pressure and heart rate will be recorded at the beginning of laryngoscopy and at the completion of intubation. Time of laryngoscopy and intubation will be recorded using a stopwatch. These data will be recorded by a second anesthesiologist who will also be taking the photograph of the glottic opening. With this technique the time to intubation will not be prolonged as a result of participating in this study.

   Even though taking a photo of glottic opening during laryngoscopy is not a routine practice we expect no significant delays in intubation or laryngoscopy.
3. Computer Editing Adobe Photoshop editing of images will be performed after collecting all data at conclusion of the study. The images will be cropped to present only the vocal cord view without the blade. The image quality and color will be approximated to ensure the images from the two different cameras (digital camera and C-MAC camera) will be similar.
4. Image grading by POGO and Cormack- Lehane scale Two anesthesiologists who are not involved in the study will be blinded to the study all together. They will review all images after they are randomized and de-identified and grade the POGO score.
5. Subjective evaluation of each blade There will be 4 anesthesiologists performing the laryngoscopies. Each patient will undergo only one laryngoscopy and tracheal intubation by one of the anesthesiologist. After the intubation, the anesthesiologist who performed the laryngoscopy and intubation will rate the difficulty of laryngoscopy and intubation on visual analogue scale 0-10 (0 representing very easy & 10 very difficult laryngoscopy/ intubation). This evaluation can be done at any time before the electronic record is completed and will not interfere with patient care.

Data Collection and Storage The investigator will use a specially designed data collection sheet. General information, demographic data, vital signs and procedure data will be recorded on this. The general information will include patient's hospital ID label, subject serial number, subject randomization group, procedure date and time. The demographic data will include age, weight, and height. The procedure data section will include the time from mask induction to IV medication administration, ease of laryngoscopy, ease of intubation and complications.

The investigators will use either a C-MAC monitor or a free standing high definition photo camera depending on the randomization group. Each photo will be saved on a SD memory card and after procedure will be transferred to Principal Investigator's computer where it will be saved under subjects serial number. At the completion of data collection of all 96 subjects the images will be edited and presented to a blinded anesthesiologist who will score each image by POGO and Cormack Lehane classification.

The data collection sheets will be kept by the principal investigator in a locked file in a locked anesthesia office. The images will be stored in principal investigator's computer that is password secured.

The data will be stored for 3 years after completion of the study by the primary investigator alone.

All data will be treated according to HIPAA practice. All collected data for this study will be de-identified for privacy protection. It will be stored using the unique study case number only, with no direct patient identifiers.

Data Analysis For the primary hypothesis of the study, the POGO scores from the Miller, Wis-Hipple size 1 blades and the C-MAC lifting the epiglottis, will be compared using the Kruskall Wallis test. For the secondary hypothesis, the POGO scores for the C-MAC 1 Miller blade lifting the epiglottis will be compared with the photos of the vocal cords taken at the lips using the Wilcoxon paired rank sum test. Data whose distribution deviate from normality (based on the Kolmogorov Smirnov test) will be presented as medians and ranges and analyzed using the above tests. Data that will be normally distributed will be presented as means and standard deviations, and analyzed using Student's t test and one-way ANOVA (with the Scheffe test) as appropriate. P < 0.05 for two tails was accepted. Data will be analyzed on an intention to treat basis.

Data Safety Monitoring Plan The safety of research participants and integrity of the data will be carefully monitored at multiple levels. The PI will be highly involved with all aspects of the protocol and will assume ultimate responsibility for the safety and well-being of research participants and the integrity of data collected. The PI will meet with each member of the study staff to ensure that they are aware of all procedures and clarify any questions they have about the protocol before initiation of the study. A record of the training sessions will be kept in the study repository. Quality control and participant safety will also be ensured via monthly supervision of research and clinical staff by PI. During these meetings the research staff will discuss the status of the research project and review the protocol, consents, any safety issues that have risen, and any additional issues to ensure that any reportable information will receive immediate and appropriate action. Each of these meetings will be documented in a log that is stored in the study repository.

ELIGIBILITY:
Inclusion Criteria:

* Children age ≤ 2 years
* American Society of Anesthesiologists (ASA) class I-II
* Fasting
* Scheduled for elective surgery under general anesthesia

Exclusion Criteria:

* Refusal by parents
* Airway surgery
* Obstructive sleep apnea
* Craniofacial abnormalities
* Predicted difficult intubation
* Prematurity < 37 gestational age
* NICU stay for > 1 week after birth
* Gastroesophageal reflux disease
* Neuromuscular disease

Ages: 1 Day to 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 96 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jerrold Lerman, MD, Principal Investigator — SUNY at Buffalo, Women and Children's Hospital of Buffalo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Passi Y, Sathyamoorthy M, Lerman J, Heard C, Marino M. Comparison of the laryngoscopy views with the size 1 Miller and Macintosh laryngoscope blades lifting the epiglottis or the base of the tongue in infants and children <2 yr of age. Br J Anaesth. 2014 Nov;113(5):869-74. doi: 10.1093/bja/aeu228. Epub 2014 Jul 25. PMID 25062740

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only 96 children had interpretable photos of the larynx: C-MAC included 36, WIs-Hipple 31 and Miller 29 children.
Pre-assignment Details: A total of 96 children were consented for the trial
Groups:
- Miller Laryngoscope Blade: A photo of the best glottic view will be taken during laryngoscopy using Miller blade. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The POGO score assesses the percent of the glottic opening that can be seen with each blade
- Wis-Hipple Laryngoscope Blade: A photo of the best glottic view will be taken during laryngoscopy using Wis- Hipple blade. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The POGO score assesses the percent of the glottic opening that can be seen with each blade
- C-Mac Laryngoscope Blade: An image of the best glottic view will be saved on C-MAC monitor's SD card during laryngoscopy using C-MAC straight blade. The view of the larynx will be assessed using the POGO score by a blinded assessor.
  Laryngoscope blade: The POGO score assesses the percent of the glottic opening that can be seen with each blade
Period: Overall Study
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade
Started | 29 | 31 | 36
Completed | 29 | 31 | 36
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade | Total
Number analyzed (Participants) | 29 | 31 | 36 | 96
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 29 | 31 | 36 | 96
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] — age in months was recorded and summarized
  months
    Age (months) | 15 (8.1) | 15 (7) | 17 (8.8) | 15 (7.35)
Sex/Gender, Customized [Number; unit: participants] — Sex/gender was NOT recorded
  participants
    Sex | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 29 | 31 | 36 | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Vocal Cord Opening
Description: The percentage of vocal cord opening (POGO) is the percent of the vocal cords that is visible during laryngoscopy. Minimum is obviously 0 and maximum 100 as in percents. The more visible the vocal cords the better the view or outcome. The mean or measure of central tendency was reported together with the 25th to 75th percentile as a measure of dispersion.
Time Frame: 10 minutes
Measure: Mean (Inter-Quartile Range); unit: percent
Groups:
- Miller Laryngoscope Blade: The percent of vocal cords (glottic opening) (POGO) score will be the estimated percent of the vocal cords visible in a photo of the larynx during laryngoscopy with a Miller laryngoscope blade in each child.
- Wis-Hipple Laryngoscope Blade: The percent of vocal cords (glottic opening) (POGO) score will be the estimated percent of the vocal cords visible in a photo of the laryngeal view during laryngoscopy with a Wish-Hipple laryngoscope blade in each child.
- C-Mac Laryngoscope Blade: The percent of vocal cord (glottic opening) (POGO) score will be the estimated percent of the vocal cords visible in a photo of the laryngeal view taken from the monitor of the C-MAC during laryngoscopy with a C-Mac laryngoscope blade and a direct view of the vocal cords using the C-Mac laryngoscope blade in each child.
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade
Number analyzed (Participants) | 29 | 31 | 36
percent | 100 [95 to 100] | 98 [92 to 100] | 100 [100 to 100]
Statistical Analysis 1: Comparison: Miller Laryngoscope Blade vs Wis-Hipple Laryngoscope Blade vs C-Mac Laryngoscope Blade; Posthoc analysis of POGO scores were compared using the Kruskall Wallis test with Mann-WHitney test for pairwise comparisons; Test type: Superiority; p < 0.05, Kruskal-Wallis

2. Secondary Outcome: Subjective Ease of Laryngoscopy and Intubation
Description: "Subjective ease of intubation" scale ranges from 1 to 10 where 1 was difficult and 10 was easy. Median and range for this nonparametric score.
Time Frame: 30 minutes from induction to tracheal intubation
Population: Median and range for the subjective ease of laryngoscopy and intubation
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade
Number analyzed (Participants) | 29 | 31 | 36
score on a scale | 10 [10 to 10] | 10 [10 to 10] | 10 [10 to 10]

3. Secondary Outcome: Percent of Oxygen Saturation
Description: percentage of oxygen saturation
Time Frame: post laryngoscopy
Measure: Median (Inter-Quartile Range); unit: percentage of oxygen saturation
Groups:
- Miller Laryngoscope Blade; Wis-Hipple Laryngoscope Blade; C-Mac Laryngoscope Blade: Oxygen saturation pre and post laryngoscopy
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade
Number analyzed (Participants) | 29 | 31 | 36
percentage of oxygen saturation | 100 [98 to 100] | 100 [99 to 100] | 100 [99 to 100]

ADVERSE EVENTS:
Time Frame: 30 minutes from induction of anesthesia until completion of tracheal intubation
Description: Definitions are the same. No adverse events occurred
Arm/Group | Miller Laryngoscope Blade | Wis-Hipple Laryngoscope Blade | C-Mac Laryngoscope Blade
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/31 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/36
Other Adverse Events (participants affected / at risk) | 0/29 | 0/31 | 0/36

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No